CLINICAL TRIAL: NCT01951651
Title: Effect of Exenatide Treatment on Myocardial Fat Content, Left Ventricular Function, and Vascular Inflammation in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Exenatide on Liver and Heart Fat and Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mandeep Bajaj, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-26030
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Glipizide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Exenatide 10 micrograms injected subcutaneously twice daily for 6 months
  Interventions: Drug: Exenatide
- Glipizide (Experimental): Glipizide 5 mg (tablet), one tablet twice daily orally for 6 months
  Interventions: Drug: Glipizide

INTERVENTIONS:
Drug: Exenatide — Type 2 diabetic subjects will be randomized to receive either Exenatide 10 micrograms twice daily injected subcutaneously or glipizide 5 mg twice daily orally for 6 months. All subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, plasma lipids, and glycosylated hemoglobin (HbA1c) as well as measurement of liver and myocardial fat content and left ventricular function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, adipocytokines, HbA1c, monocyte inflammation, as well as hepatic/myocardial fat content determination and left ventricular function at the end of the 6 months.
  Other Names: Byetta
  Arms: Exenatide
Drug: Glipizide — Type 2 diabetic subjects will be randomized to receive either Exenatide 10 micrograms twice daily injected subcutaneously or glipizide 5 mg twice daily orally for 6 months. All subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, plasma lipids, and glycosylated hemoglobin (HbA1c) as well as measurement of liver and myocardial fat content and left ventricular function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, adipocytokines, HbA1c, monocyte inflammation, as well as hepatic/myocardial fat content determination and left ventricular function at the end of the 6 months.
  Other Names: Glucotrol
  Arms: Glipizide

SUMMARY:
The purpose of this study is to examine the effect of exenatide on liver and heart (myocardial) fat and inflammation.

DETAILED DESCRIPTION:
Type 2 diabetics and insulin resistant individuals have an excess of fat in the liver which is not attributable to alcohol or other known causes of liver disease, a condition defined as nonalcoholic fatty liver disease (NAFLD). The fatty liver is insulin resistant. Individuals with a fatty liver are more likely to have excess intra-abdominal fat as well as a reduction in circulating plasma adiponectin levels. We have previously shown that type 2 diabetes and its associated Non Alcoholic Fatty Liver Disease (NAFLD) is characterized by increased hepatic fat content, decreased circulating adiponectin levels, and hepatic and peripheral (muscle) insulin resistance. Weight loss in humans with Non Alcoholic Fatty Liver Disease is associated with a decrease in hepatic fat content. Exenatide, an incretin based anti-diabetes therapy, enhances glucose-dependent insulin secretion and glucose-dependent suppression of inappropriately high glucagon secretion, improves glycemic control in patients with type 2 diabetes and is associated with weight loss. In rodent studies, exenatide reduces hepatic and myocardial fat and reduces vascular inflammation independent of changes in weight. Exenatide has also been shown to increase plasma adiponectin levels in humans and rodents. Furthermore type 2 diabetics are characterized by an increase in both hepatic and myocardial fat and left ventricular dysfunction, particularly diastolic dysfunction. However, the effect of exenatide therapy on liver and myocardial fat content, as well as left ventricular function in patients with type 2 diabetes has not been previously studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Patients may be of either sex. Female patients must be non-lactating and must either be at least two years post-menopausal, or be using adequate contraceptive precautions.
3. Patients must range in age from 30 to 70 years, inclusive.
4. Patients must meet the American Diabetes Association (ADA) criteria (ADA 1997 Criteria: fasting plasma glucose greater than or equal to 126 mg/dl) for the diagnosis of type 2 diabetes mellitus.
5. Patients must be on diet therapy and/or metformin treatment for type 2 diabetes (stable dose)and have a fasting plasma glucose concentration between 126 and 260 mg/dl
6. Patients must have Hematocrit greater than 34 vol%.
7. Subjects whose body weight has been stable over the three months prior to study enrollment will be included.

Exclusion Criteria:

1. Patients must not have type 1 diabetes.
2. Patients must not have a fasting plasma glucose greater than 260 mg/dl.
3. Patients must not have received a thiazolidinedione for at least 3 months prior to randomization.
4. Patients must not be on insulin treatment or have received insulin for more than one week within the previous year prior to entry. Patients should not be on sulfonylureas, sitagliptin, or exenatide treatment.
5. Patients taking systemic glucocorticoids or other medications known to affect glucose tolerance are excluded.
6. Patients taking medications that affect gastrointestinal motility will be excluded.
7. Patients with a history of Congestive Heart Failure, or clinically significant cardiac, liver or kidney disease (creatinine greater than 1.5 mg/dl).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Bajaj, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide | Glipizide
Started | 12 | 12
Completed | 8 | 10
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Glipizide | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Fat Content
Description: Myocardial fat content following intervention as measured by magnetic resonance imaging and spectroscopy (MRS) in patients with type 2 diabetes.
Time Frame: 6 months
Population: One patient assigned to the glipizide treatment arm did not complete the myocardial fat content study (MRS) following 6 months of treatment
Measure: Mean (Standard Error); unit: percentage of myocardium content
Arm/Group | Exenatide | Glipizide
Number analyzed (Participants) | 8 | 9
percentage of myocardium content | 1.7 (0.4) | 1.1 (0.2)

2. Primary Outcome: Hepatic Fat Content
Description: Hepatic fat content following intervention in patients with type 2 diabetes
Time Frame: 6 months
Population: One patient assigned to the glipizide treatment arm did not complete the hepatic fat content study (MRS) following 6 months of treatment
Measure: Mean (Standard Error); unit: percent of hepatic fat
Arm/Group | Exenatide | Glipizide
Number analyzed (Participants) | 8 | 9
percent of hepatic fat | 10.9 (1.8) | 13.1 (3.5)

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)(%).
Description: Left Ventricular Ejection Fraction following intervention as measured by magnetic resonance imaging in patients with type 2 diabetes.
Time Frame: 6 months
Population: One patient assigned to the glipizide treatment arm did not complete the Left Ventricular Ejection Fraction study (magnetic resonance imaging) following 6 months of treatment
Measure: Mean (Standard Error); unit: percent of Left ventricular function
Arm/Group | Exenatide | Glipizide
Number analyzed (Participants) | 8 | 9
percent of Left ventricular function | 60 (5) | 56 (2)

4. Secondary Outcome: Monocyte Inflammatory Protein Nuclear Factor Kappa-B (NFkappaB) (%)
Description: The percentage change in monocyte inflammatory proteins NFkappaB (%) from baseline.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Exenatide | Glipizide
Number analyzed (Participants) | 8 | 10
percentage change from baseline | -65.0 (8.0) | 0.0 (3.0)

ADVERSE EVENTS:
Arm/Group | Exenatide | Glipizide
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes